CLINICAL TRIAL: NCT01440192
Title: A Phase 1B, Multi-Center, Open-Label, Single Dose Study to Evaluate the Safety of Intravenous Infusion of Human Placental-Derived Cells (PDA001) for the Treatment of Adults With Stage II or III Pulmonary Sarcoidosis.Sarcoidosis
Brief Title: Safety of Intravenous Infusion of Human Placenta-Derived Cells (PDA001) for the Treatment of Adults With Stage II or III Pulmonary Sarcoidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Terminated by Sponsor
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT-PDA001-SAR-001
Record Dates: First submitted 2011-09-19; First posted 2011-09-26 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2014-07

CONDITIONS: Stage 2 Pulmonary Sarcoidosis; Stage 3 Pulmonary Sarcoidosis
Keywords: Sarcoidosis; Stem cells; PDA001; Celgene; Human Placenta-Derived cells; Cenplacel-L
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A: 1 Unit PDA001 (cenplacel-L) (Experimental)
  Interventions: Biological: PDA001 (cenplacel-L)
- Cohort B: 1 Unit PDA001 (cenplacel-L) (Experimental): 1 unit PDA001(cenplacel-L)
  Interventions: Biological: PDA001 (cenplacel-L)

INTERVENTIONS:
Biological: PDA001 (cenplacel-L) — 1 unit PDA001 (approximately 200 x 106 cells) IV on Days 1 & 8
  Other Names: Human Placenta-Derived Cells

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of a single dose of PDA001 (given twice) in subjects with Stage II or III Pulmonary Sarcoidosis (PS) who are refractory to one or more of the following treatments for PS: methotrexate,immunosuppressants or cytotoxic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years to 75 years of age at the time of signing the informed consent document
2. Understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures are conducted
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. Weight must be ≥ 50 kg
5. A female of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 24 hours prior to treatment with study therapy. In addition, sexually active FCBP must agree to use two of the following adequate forms of contraception methods simultaneously such as: oral, injectable or implantable hormonal contraception; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner for the duration of the study and the follow-up period. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP for the duration of the study and the follow-up period
6. Diagnosis of sarcoidosis as evidenced by parenchymal disease on chest radiograph (Stage II or III), as well as histologic confirmation of granulomatous inflammation and disease duration of ≥ 1 year
7. Refractory to one or more of the following; methotrexate, immunosuppressants or cytotoxic agents
8. Forced vital capacity (FVC) of ≥ 45% and ≤ 80% of predicted normal value at screening
9. Must be on a stable dose of prednisone, methotrexate, and/or azathioprine for pulmonary Sarcoidosis for 4 weeks prior to infusion of the IP

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
2. Any condition that confounds the ability to interpret data from the study
3. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
4. Subjects with Stage I or Stage IV sarcoidosis
5. Subjects with cutaneous sarcoidosis only
6. Subjects with neurosarcoidosis or (clinically apparent) cardiac sarcoidosis
7. Lung disease, other than sarcoid related, such as asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD)
8. History of listeriosis, coccidiomycosis, histoplasmosis, blastomycosis, treated or untreated tuberculosis or exposure to individuals with tuberculosis
9. History of pulmonary emboli or deep vein thrombus
10. Active smoker or previous smoker > 10 pack years (PY). Previous smokers must have discontinued smoking for at least 1 year
11. Morbidly obese [Body Mass Index (BMI)] > 35 at screening)
12. Inability to perform 6 Minute Walk Test (6MWT) or Pulmonary Function Test (PFT) maneuvers
13. Sickle cell disease (Hemoglobin SS, Hemoglobin SC, and sickle cell-beta thalassemia)
14. Treatment at any time with B cell depleting therapies
15. Any biologic anti-tumor necrosis factor (anti-TNF) therapy within the previous year
16. Active infection requiring treatment within 30 days prior to screening
17. Pregnant or lactating females
18. Aspartate transaminase (AST), alanine aminotransferase (ALT) or creatine phosphokinase (CPK) > 2 x the upper limit of normal at screening
19. Active infection with hepatitis B or hepatitis C
20. Known infection with human immunodeficiency virus (HIV)
21. Creatinine level > 1.5 times the upper limit of normal
22. Platelet count < 100,000/µL (< 100 x 109/L)
23. White blood cell count < 3,000/cu mm (< 3.0 x 109/L) or >20,000/cu mm (> 20 x 109/L)
24. Organic heart disease (e.g., congestive heart failure, cor pulmonale), myocardial infarction within six months prior to screening
25. Clinically significant findings on electrocardiogram (ECG) at screening (eg, arrhythmia)
26. History of other malignancies within 5 years (except basal cell carcinoma of the skin that is surgically cured, remote history of cancer now considered cured or positive Pap smear with subsequent negative follow-up)
27. Documented prior history of neurological disease or evidence of ongoing neurological disease
28. Known allergy to bovine or porcine products
29. Subject has received an investigational agent (an agent or device not approved by Federal Drug Administration (FDA) for marketed use in any indication) within 90 days (or 5 half-lives, whichever is longer) prior to treatment with investigational product (IP)
30. Subject who has received previous cell therapy
31. Subject is expecting to have elective surgery within 12 weeks prior to or post dosing with IP if the surgery would be expected to confound evaluation of outcome endpoints

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Evaluate pulmonary artery pressure during infusion | Day 1
  Evaluate pulmonary artery pressure during infusion
Adverse Events | 24 months ( 2 years) from first dose - Study Day 1
  Number of Participants experiencing adverse events during the initial and extended follow-up periods
Evaluate pulse oximetry during infusion | Day 1 and Day 8
  Evaluate pulse oximetry during infusion on Day 1 and on Day 8.

SECONDARY OUTCOMES:
Change from baseline thru study day 731 in forced vital capacity (FVC) | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in forced vital capacity (FVC)
Change from baseline thru study day 731 in forced expiratory volume (FEV1) | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in forced expiratory volume (FEV1)
Change from baseline thru study day 731 in diffusing capacity of the lung for carbon monoxide (DLCO) | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in diffusing capacity of the lung for carbon monoxide (DLCO)
Change from baseline thru study day 731 in 6 minute walk test (6MWT) | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in 6 minute walk test (6MWT)
Change from baseline thru study day 731 in St. George's Respiratory Questionnaire (SGRQ). | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in St. George's Respiratory Questionnaire (SGRQ).
Change from baseline thru study day 731 in Fatigue Assessment Score (FAS) | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in Fatigue Assessment Score (FAS)
Change from baseline thru study day 731 in baseline dyspnea index (BDI)/ transitional dyspnea index (TBI | 24 months ( 2 years) from first dose - Study Day 1
  Change from baseline thru study day 731 in baseline dyspnea index (BDI)/ transitional dyspnea index (TBI

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Luchi, MD, Study Director — Celularity Incorporated
Locations (4):
- United States (4):
  - University of Alabama, Birmingham - Division of Pulmonary, Allergy, and Critical Care Medicine, Birmingham, Alabama
  - National Jewish Health, Denver, Colorado
  - University of Cincinatti Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation - Respiratory Institute, Cleveland, Ohio